CLINICAL TRIAL: NCT02467231
Title: Ovarian Reserve After Cancer: Longitudinal Effects A Multicenter Prospective Cohort Study by the Oncofertility Consortium
Brief Title: Ovarian Reserve After Cancer: Longitudinal Effects
Acronym: ORACLE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 809406
Record Dates: First submitted 2013-07-22; First posted 2015-06-09 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Effects of Chemotherapy; Premature Ovarian Failure
Keywords: new diagnosis of cancer; chemotherapy; oncofertility; alkylating agent; fertility preservation; fertility after cancer; late effects
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exposed: Females ages 11-35 to be exposed to alkylating agent chemotherapy

SUMMARY:
Women of reproductive age who will receive treatment for cancer that includes chemotherapy may participate in a study measuring ovarian function over time. Eligible women are asked to complete a questionnaire, a menstrual diary, a brief physical examination, an ultrasound, and a blood test before, during and after cancer treatment.

DETAILED DESCRIPTION:
A total of 7 study visits will be completed at 3 month intervals including 1 visit prior to treatment, and at least 2 visits after completion of treatment. Duration of study participation is 18-30 months, depending on length of treatment.

Review and Documentation of Cancer Therapy will be abstracted from the clinical oncology chart by the oncology offices caring for the patient. Treatment will be summarized in terms of chemotherapeutic type, duration and cumulative dose; total radiation dose and location; history and type of bone marrow transplantation; and any surgery. Any attempts at fertility preservation or use of gonadotropin releasing hormone agonist treatment during cancer therapy will be captured as well.

ELIGIBILITY:
Inclusion Criteria for exposed population:

* Postmenarchal females to be treated with chemotherapy
* between the ages of 11-35 years,
* with a uterus and at least one ovary

Inclusion Criteria for unexposed population:

* healthy postmenarchal females
* no prior or planned exposure to chemotherapy
* between the ages of 11-35,
* with a uterus and at least one ovary
* regular menstrual cycles (21-35 days)

Exclusion criteria for all subjects:

* positive pregnancy test at enrollment
* lactation within the previous 1 month,
* previous treatment with chemotherapy or radiation therapy with the exception of radioactive iodine for thyroid cancer.
* previous diagnosis of an illness associated with premature ovarian failure (Turner's syndrome, Fragile X permutation carrier)
* endocrine disorder associated with irregular menstrual cycles (Cushing's disease, Thyroid disease, hyper-prolactinemia, congenital adrenal hyperplasia).

Additional exclusions for the unexposed population:

* a history of infertility, defined as at least 12 months of unprotected intercourse without conception
* polycystic ovary syndrome (PCOS)

Ages: 11 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Postmenarchal females, ages 11-35, who will require chemotherapy; An unexposed cohort balanced to the exposed cohort with respect to age and oral contraceptive use.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2009-02; Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in reproductive hormone measures, during and after chemotherapy. | 18-30 months: pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  20 mls blood will be obtained at stated timepoints for determining levels of Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2), Inhibin B, and Anti-mullerian Hormone (AMH). In menstruating girls and young women hormone measures will be obtained during the early follicular phase of the menstrual cycle (days 1-4). In women with irregular cycles the testing will be done spontaneously without regard for the bleeding pattern.

SECONDARY OUTCOMES:
Change from baseline in antral follicle counts, during and after chemotherapy. | 18-30 months: pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  All ovarian follicles and cysts will be measured by transvaginal or transabdominal ultrasound. Follicles will be measured in millimeters and grouped according to size: 2-5 mm, 6-9 mm, and >10 mm in diameter.

OTHER OUTCOMES:
Change from baseline in menstrual function, during and after chemotherapy | 18-30 months: Pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  Subjects are asked to document menstrual bleeding in a diary, noting duration of each menstrual period in days, bleeding intensity (spotting, light, moderate, heavy, flooding, none), and intervals between periods.
Change from baseline in menopausal symptoms during and after chemotherapy. | 18-30 months: Pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  The validated "Menopausal Symptom List" (MSL) will be used at each study visit to assess the presence or absence of menopausal symptoms during the past month, the frequency and severity of each symptom. Symptoms captured include: hot flashes, vaginal dryness, concentration/memory problems, irritability, mood swings, feeling sad, feeling anxious, trouble sleeping, aches, joint pain, headaches.
Change from baseline in ovarian volume during and after chemotherapy. | 18-30 months: Pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  Ovaries will be measured in three dimensions. Uterine size and endometrial thickness will also be performed. The transvaginal approach is preferred, but transabdominal ultrasound will be performed in girls who do not feel comfortable with the transvaginal procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Clarisa R Gracia, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Reproductive Research Unit, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Dillon KE, Sammel MD, Prewitt M, Ginsberg JP, Walker D, Mersereau JE, Gosiengfiao Y, Gracia CR. Pretreatment antimullerian hormone levels determine rate of posttherapy ovarian reserve recovery: acute changes in ovarian reserve during and after chemotherapy. Fertil Steril. 2013 Feb;99(2):477-83. doi: 10.1016/j.fertnstert.2012.09.039. Epub 2012 Oct 18. PMID 23084267
- [Derived] Cameron K, Sammel MD, Prewitt M, Gracia C. Differential Rates of Change in Measures of Ovarian Reserve in Young Cancer Survivors Across the Reproductive Lifespan. J Clin Endocrinol Metab. 2019 May 1;104(5):1813-1822. doi: 10.1210/jc.2018-02257. PMID 30566616